CLINICAL TRIAL: NCT00791154
Title: QUILT-2.013 A Phase 1b/2 Trial of AMG 479 or AMG 102 in Combination With Platinum-based Chemotherapy as First-Line Treatment for Extensive Stage Small Cell Lung Cancer
Brief Title: QUILT-2.013: First-Line Treatment for Extensive Stage Small Cell Lung Cancer
Acronym: SCLC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Subjects discontinued study
Sponsor: NantCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QUILT-2.013; NCT00791154 (Other: NantCell)
Record Dates: First submitted 2008-10-23; First posted 2008-11-14 (Estimated); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Lung Cancer; Small Cell Lung Cancer; Solid Tumors; Extensive-stage Small Cell Lung Cancer
Keywords: Extensive disease; Extrathoracic metasasis; Malignant pericardial effusion; Malignant pleural effusion; Contralateral hilar adenopathy
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma; Pleural Effusion, Malignant | interventions — ganitumab; Etoposide; rilotumumab; Carboplatin; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- ARM A (Experimental): Blinded AMG 479 study drug and carboplatin or cisplatin and etoposide
  Interventions: Drug: AMG 479; Drug: Etoposide; Drug: Carboplatin; Drug: Cisplatin
- ARM B (Experimental): Blinded AMG 102 study drug and carboplatin or cisplatin and etoposide
  Interventions: Drug: Etoposide; Drug: AMG 102; Drug: Carboplatin; Drug: Cisplatin
- ARM C (Placebo Comparator): Blinded placebo and carboplatin or cisplatin and etoposide
  Interventions: Drug: Etoposide; Drug: Placebo; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Drug: AMG 479 — AMG 479 is administered to subjects
  Arms: ARM A
Drug: Etoposide — Etoposide is administered to subjects
Drug: Placebo — Placebo is administered with Carboplatin and Etoposide
  Arms: ARM C
Drug: AMG 102 — AMG 102 is administered to subjects
  Arms: ARM B
Drug: Carboplatin — Carboplatin is administered to some subjects in combination
Drug: Cisplatin — Cisplatin is administered to some subjects in combination

SUMMARY:
This trial is titled "A Phase 1b/2 trial of AMG 479 or AMG 102 with Platinum-Based Chemotherapy as First-Line Treatment for Extensive Stage Small-Cell Lung Cancer (SCLC)."

Part 1, the phase 1b portion of this study, is a multicenter, open-label investigation to identify safe dose levels of either AMG 102 or AMG 479 in combination with etoposide plus cisplatin or carboplatin in subjects with previously untreated extensive stage SCLC.

Part 2, the phase 2 portion of this study, is a multicenter, double-blind, 3-arm investigation to evaluate overall survival of either AMG 102 or AMG 479 in combination with platinum-based chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria

* Histologically or cytologically confirmed SCLC
* Extensive disease, defined by at least one of the following:
* No limited disease (ie, no disease confined to the ipsilateral hemithorax, which can be safely encompassed within a tolerable radiation field)
* Extrathoracic metastases
* Malignant pericardial or pleural effusion
* Contralateral hilar adenopathy
* Measurable or nonmeasurable disease, as defined by modified RECIST
* Eastern Cooperative Oncology Group (ECOG) status 0 or 1
* ≥18 years old
* Life expectancy (with therapy) ≥3 months
* Adequate hematologic, hepatic, coagulation, renal, and metabolic function
* Diabetes, if present, must be controlled, with glycosylated hemoglobin (HbA1C) ≤ 8% and fasting glucose levels ≤160 mg/dL

Key Exclusion Criteria

* Prior chemotherapy, chemoradiation, or investigational agent for SCLC
* Prior radiotherapy to >25% of the bone marrow
* Symptomatic or untreated central nervous system metastases (with exceptions)
* Currently or previously treated with biologic, immunologic or other therapies for SCLC
* Current serious or nonhealing wound or ulcer
* History of prior concurrent other malignancy (with exceptions)
* Thorombosis or vascular ischemic events within the last 12 months such as DVT, PE, TIA or MI
* Any clinically significant medical condition other than cancer (eg, cardiovascular disease or COPD), which could interfere with the safe delivery of study treatment or risk of toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2008-12-02 (Actual); Primary Completion 2010-02-02 (Actual); Study Completion 2013-05-01 (Actual)

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: AMG 479/Carboplatin+Etoposide: AMG 479 in combination with etoposide plus carboplatin (Cohort 1)
- Phase 1: AMG 479/Cisplatin+Etoposide: cisplatin (Cohort 2)
- Phase 1: AMG102/Carboplatin+Etoposide: AMG 102 in combination with etoposide plus carboplatin (Cohort 3)
- Phase 1: AMG 102/Cisplatin+Etoposide: cisplatin (Cohort 4)
- Phase 2 Ganitumab: Blinded AMG 479 study drug and carboplatin or cisplatin and etoposide
- Phase 2 Rilotumumab: Blinded AMG 102 study drug and carboplatin or cisplatin and etoposide
- Phase 2 Placebo: Blinded placebo and carboplatin or cisplatin and etoposide
Period: Overall Study
Arm/Group | Phase 1: AMG 479/Carboplatin+Etoposide | Phase 1: AMG 479/Cisplatin+Etoposide | Phase 1: AMG102/Carboplatin+Etoposide | Phase 1: AMG 102/Cisplatin+Etoposide | Phase 2 Ganitumab | Phase 2 Rilotumumab | Phase 2 Placebo
Started | 6 | 8 | 6 | 8 | 62 | 62 | 61
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 8 | 6 | 8 | 62 | 62 | 61
Not completed — Noncompliance | 0 | 1 | 0 | 0 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Full Consent withdrawn | 1 | 3 | 0 | 0 | 1 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 2 | 0 | 4
Not completed — Death | 5 | 4 | 4 | 7 | 54 | 54 | 52
Not completed — Other event | 0 | 0 | 2 | 0 | 2 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: AMG 479/Carboplatin+Etoposide | Phase 1: AMG 479/Cisplatin+Etoposide | Phase 1: AMG102/Carboplatin+Etoposide | Phase 1: AMG 102/Cisplatin+Etoposide | Phase 2 Ganitumab | Phase 2 Rilotumumab | Phase 2 Placebo | Total
Number analyzed (Participants) | 6 | 8 | 6 | 8 | 62 | 62 | 61 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (7.3) | 55.4 (9.0) | 60.7 (8.0) | 59.4 (5.0) | 59.8 (7.6) | 60.8 (7.6) | 59.6 (9.7) | 60.1 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 2 | 14 | 15 | 14 | 54
  Male | 2 | 6 | 3 | 6 | 48 | 47 | 47 | 159
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 4 | 1 | 1 | 13 | 13 | 6 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 4 | 5 | 7 | 48 | 49 | 55 | 174
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Histologically or cytologically confirmed SCLC [Count of Participants; unit: Participants] | 6 | 7 | 6 | 8 | 62 | 62 | 61 | 212

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival in Ganitumab Treated Subjects -Phase 2
Description: The primary efficacy endpoint was overall survival, defined as time from randomization to death from any cause
Time Frame: Time from randomization to death from any cause, approximately 14 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Ganitumab | Phase 2 Placebo
Number analyzed (Participants) | 62 | 61
months | 10.7 [8.1 to 14.1] | 10.8 [9.4 to 11.9]

2. Primary Outcome: Overall Survival in Rilotumumab Treated Subjects-Phase 2
Description: The primary efficacy endpoint is overall survival, defined as time from randomization to death from any cause
Time Frame: Time from randomization to death from any cause, approximately 14 months
Population: This endpoint was phase 2 subjects only
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 1: AMG 102/Cisplatin+Etoposide: AMG 102 in combination with etoposide plus carboplatin (Cohort 3) or cisplatin (Cohort 4)
Arm/Group | Phase 1: AMG 479/Carboplatin+Etoposide | Phase 1: AMG 479/Cisplatin+Etoposide | Phase 1: AMG102/Carboplatin+Etoposide | Phase 1: AMG 102/Cisplatin+Etoposide | Phase 2 Rilotumumab | Phase 2 Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 62 | 61
months |  |  |  |  | 12.2 [8.8 to 14.6] | 10.8 [9.4 to 11.9]

3. Primary Outcome: Number of Subjects With Dose Limiting Toxicities-Phase 1
Description: For Part 1, DLTs were defined as the incidence during the first 21 days of starting study treatment of any Grade 3 or higher hematologic or non-hematologic toxicity related to AMG 479 or AMG 102, or the combination of AMG 479 or AMG 102 with chemotherapy, except for lymphocytopenia and anemia. DLTs did not include fatigue, nausea, diarrhea, vomiting, hyperglycemia, neutropenia, thrombocytopenia, increased AST or ALT, or pulmonary embolism unless specific criteria were met as stated in protocol section 6.1.3.2.
Time Frame: First 21 days after start of study treatment
Population: This endpoint is for phase 1 subjects only
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: AMG 479/Carboplatin+Etoposide | Phase 1: AMG 479/Cisplatin+Etoposide | Phase 1: AMG102/Carboplatin+Etoposide | Phase 1: AMG 102/Cisplatin+Etoposide | Phase 2 Ganitumab | Phase 2 Rilotumumab | Phase 2 Placebo
Number analyzed (Participants) | 6 | 7 | 6 | 8 | 0 | 0 | 0
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All serious adverse events that occur after the subject has signed the informed consent form through to the Safety Follow-up Visit or 30 days after completion of the study treatment phase, approximately 14 months. All non-serious adverse events that occur after the subject has enrolled through to the Safety Follow-up Visit or 30 days after completion of the study treatment phase, approximately 14 months.
Description: The Safety population was used for adverse event reporting (i.e., all subjects that had at least one dose of study drug). All subjects were measured for mortality.
Groups:
- Phase 1: AMG 479/Carboplatin+Etoposide: combination with etoposide plus carboplatin (Cohort 1)
- Phase 1: AMG 479/Cisplatin+Etoposide: Phase 1: AMG 479/Cisplatin+Etoposide cisplatin (Cohort 2)
- Phase 1: AMG 102/Cisplatin+Etoposide: Phase 1: AMG 102/Cisplatin+Etoposide cisplatin (Cohort 4)
Arm/Group | Phase 1: AMG 479/Carboplatin+Etoposide | Phase 1: AMG 479/Cisplatin+Etoposide | Phase 1: AMG102/Carboplatin+Etoposide | Phase 1: AMG 102/Cisplatin+Etoposide | Phase 2 Ganitumab | Phase 2 Rilotumumab | Phase 2 Placebo
All-Cause Mortality (participants affected / at risk) | 5/6 | 4/8 | 4/6 | 7/8 | 54/62 | 54/62 | 52/61
Serious Adverse Events (participants affected / at risk) | 5/6 | 2/7 | 4/6 | 7/8 | 7/59 | 6/61 | 3/59
Other Adverse Events (participants affected / at risk) | 6/6 | 6/7 | 6/6 | 8/8 | 58/59 | 61/61 | 57/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: AMG 479/Carboplatin+Etoposide (N=6) | Phase 1: AMG 479/Cisplatin+Etoposide (N=7) | Phase 1: AMG102/Carboplatin+Etoposide (N=6) | Phase 1: AMG 102/Cisplatin+Etoposide (N=8) | Phase 2 Ganitumab (N=59) | Phase 2 Rilotumumab (N=61) | Phase 2 Placebo (N=59)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Septic Shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Septic Embolus (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Septic Shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Medication Error (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Superior Vena Cava Syndrome (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Venous Thrombosis Limb (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: AMG 479/Carboplatin+Etoposide (N=6) | Phase 1: AMG 479/Cisplatin+Etoposide (N=7) | Phase 1: AMG102/Carboplatin+Etoposide (N=6) | Phase 1: AMG 102/Cisplatin+Etoposide (N=8) | Phase 2 Ganitumab (N=59) | Phase 2 Rilotumumab (N=61) | Phase 2 Placebo (N=59)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 24 | 18 | 13
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 13 | 8 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 24 | 14 | 16
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 11 | 6 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 13 | 8 | 7
Weight Decreased (Investigations) | 0 | 0 | 0 | 0 | 7 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 5 | 12 | 10
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 15 | 11 | 10
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 16 | 7 | 11
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 15 | 15 | 10
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 6 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 13 | 8 | 9
Hyperglycaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 5 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 0
Back Pain (General disorders) | 0 | 0 | 0 | 0 | 4 | 5 | 7
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 5 | 0 | 2
Oropharyngeal Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 5
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Hypokalaemia (Investigations) | 0 | 0 | 0 | 0 | 3 | 6 | 0
Ototoxicity (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1 | 3 | 3 | 0 | 0
Headache (General disorders) | 0 | 0 | 0 | 0 | 8 | 5 | 5
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 1 | 5 | 5 | 8
Hyponatraemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 5
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 5 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 6 | 3 | 7
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 8 | 6 | 9
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 7 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 4 | 5 | 5 | 41 | 36 | 42
Oedema Peripheral (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 8 | 2
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 3 | 4 | 0 | 0 | 0
Anaemia Macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobinaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1 | 2 | 2 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry Eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye Pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid Disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eyelid Oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphthous Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Chapped Lips (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 3 | 1 | 3 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 2 | 3 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Gingival Bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 3 | 5 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral Disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2 | 2 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 1 | 3 | 4 | 0 | 0 | 0
Catheter Site Inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest Discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Face Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 4 | 0 | 0 | 0 | 0
Infusion Site Extravasation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal Inflammation (General disorders) | 2 | 1 | 2 | 1 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0
Pyrexia (General disorders) | 4 | 1 | 2 | 1 | 0 | 0 | 0
Cytolytic Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Balanitis Candida (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis Bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral Fungal Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 2 | 0 | 1 | 2 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Septic Embolus (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Septic Shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Medication Error (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood Creatinine Increased (Investigations) | 1 | 1 | 0 | 2 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Brain Natriuretic Peptide Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glomerular Filtration Rate Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet Count Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Troponin Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Troponin T Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 1 | 1 | 4 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 1 | 1 | 4 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight Fluctuation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 2 | 0 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysgraphia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Formication (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 2 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Memory Impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Reproductive system and breast disorders) | 1 | 2 | 2 | 3 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4 | 0 | 0 | 0
Pulmonary Thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sputum Discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 4 | 3 | 5 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 2 | 1 | 0 | 0 | 0
Superior Vena Cava Syndrome (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Venous Thrombosis Limb (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-04-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT00791154/Prot_SAP_000.pdf